CLINICAL TRIAL: NCT03334110
Title: Clinical Randomized Controlled Trial of the New Method of Selective Coronary Venous Bypass Graft on Improving Curative Effects in Patients With Diffuse Coronary Artery Disease
Brief Title: A Clinical Randomized Controlled Trial of the New Method of Selective Coronary Vein Bypass Graft (SCVBG)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yang Yu, Professor；Chief Physician；, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Z151100004015177
Record Dates: First submitted 2017-09-17; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Coronary Atherosclerotic Heart Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIMA-GSV-SCVBG Group (Experimental): Experimental group: The intervention：we apply a new operation on the patients with diffuse coronary artery disease(DCAD), we choose LIMA-GSV composited Y graft and anastomose the GSV with selective coronary vein.
  Interventions: Procedure: A method of operation: LIMA-GSV-SCVBG
- BIMA-SCVBG Group (Other): The other group：The intervention: We choose bilateral internal mammary artery composited LIMA-Right Mammary Internal Artery（RIMA） y graft， and anastomose the RIMA with selective coronary vein.
  Interventions: Procedure: BIMA-SCVBG

INTERVENTIONS:
Procedure: A method of operation: LIMA-GSV-SCVBG — On the experimental group,We treat patients with the operation of LIMA-GSV composited Y graft and anastomose the GSV with selective coronary vein
  Arms: LIMA-GSV-SCVBG Group
Procedure: BIMA-SCVBG — On the other group, We treat patients with the operation of bilateral internal mammary artery composited LIMA-Right Mammary Artery（RIMA） y graft and anastomose the Right Mammary Artery(RIMA) with selective coronary vein.
  Arms: BIMA-SCVBG Group

SUMMARY:
Apply a new operation method of Left Internal Mammary Artery (LIMA)-Greater Saphenous Vein (GSV)-SCVBG to the treatment of patients with diffuse coronary artery disease,through clinical randomized controlled study,compared with patients of bilateral internal mammary artery (BIMA)-SCVBG and evaluate both of therapeutic effects and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with right coronary artery diffuse lesions:Right coronary artery lumen≤1mm，Lesion lengths ≥20mm or multiple segment lesions.
* Patients of coronary artery bypass grafting (CABG) that can't be treated through endarterectomy.
* Patients ≤ 70 years old.
* All enrolled patients must being signed the informed consent.

Exclusion Criteria:

* Severe heart failure(ejection fraction under 35%) or non coronary atherosclerotic heart disease patients such as combined with severe valvular heart disease.
* Patients with acute myocardial infarction.
* Assistant examinations indicate that the bridge vessels can't be used；The left subclavian artery stenosis and/or LIMA lesions；RIMA lesions；varicosis of both great saphenous vein.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2017-11-30 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
The patency rate of bridge vessels and selective coronary vein | 1-3 years
  We will assess the patency rate during a follow-up of 1 year, and continue to follow up to 3 years after the end of the project

SECONDARY OUTCOMES:
Main adverse cardiovascular and cerebrovascular events | 1-3 years
  We will follow up the main adverse cardiovascular and cerebrovascular events ( death, myocardial infarction, stroke and repeated revascularization) 7 days, 1 month, 3 months, 6 months and 1 year after the operation and continue to 3 years.
Wound complications | 1-3 years
  We will follow up the wound complications (sternum and mediastinal infection, incision infection, fat liquefaction) 7 days, 1 month, 3 months, 6 months and 1 year after the operation and continue to 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing An Zhen Hospital , Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided